CLINICAL TRIAL: NCT00725075
Title: A Multi-center, Double-blind, Flexible-dose Efficacy Trial With Org 25935 Versus Placebo as add-on Therapy in Subjects With Predominant, Persistent Negative Symptoms of Schizophrenia Treated With a Stable Dose of a Second Generation Antipsychotic (GIANT)
Brief Title: Adjuvant Treatment With a Glycine Uptake Inhibitor in Participants With Negative Symptoms of Schizophrenia (P05695) (MK-8435-001)
Acronym: GIANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05695; MK-8435-001 (Other: Merck Registration Number); 172003 (Other: Organon Protocol Number); P05695 (Other: Schering-Plough Protocol Number); 2006-003080-31 (EudraCT Number)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Schizophrenia
Keywords: Negative symptoms; Glycine Uptake inhibitor; Add-on treatment; Second Generation Antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — N-methyl-N-(6-methoxy-1-phenyl-1,2,3,4-tetrahydronaphthalen-2-ylmethyl)aminomethylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MK-8435 (Org 25935) 8-16 mg per day (Experimental): Participants will be maintained on a stable dose of Second Generation Antipsychotic (SGA) and receive 4-8 mg MK-8435 (Org 25935) BID, in the morning and the evening, as add-on treatment for up to 87 days. The dose of MK-8435 (Org 25935) can be titrated upward or downward within the specified dose range, as needed, up to Day 42 of the study. The dose must remain stable after Day 42 for the remainder of the study.
  Interventions: Drug: MK-8435 (Org 25935) 4-8 mg
- MK-8435 (Org 25935) 24-32 mg per day (Experimental): Participants will be maintained on a stable dose of SGA and receive 12-16 mg MK-8435 (Org 25935) BID, in the morning and the evening, as add-on treatment for up to 87 days. The dose of MK-8435 (Org 25935) can be titrated upward or downward within the specified dose range, as needed, up to Day 42 of the study. The dose must remain stable after Day 42 for the remainder of the study.
  Interventions: Drug: MK-8435 (Org 25935) 12-16 mg
- Placebo (Placebo Comparator): Participants will be maintained on a stable dose of SGA and receive matching placebo for MK-8435 (Org 25935) BID, in the morning and the evening, as add-on treatment for up to 87 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8435 (Org 25935) 4-8 mg — Administered orally 2 times a day (BID) for a final concentration of 8-16 mg/day
  Arms: MK-8435 (Org 25935) 8-16 mg per day
Drug: Placebo — Matching placebo for MK-8435 (Org 25935) administered orally BID
  Arms: Placebo
Drug: MK-8435 (Org 25935) 12-16 mg — Administered orally BID for a final concentration of 24-32 mg/day
  Arms: MK-8435 (Org 25935) 24-32 mg per day

SUMMARY:
The purpose of this study is to determine whether MK-8435 (Org 25935) is more effective than placebo in improving negative symptoms in participants with schizophrenia who are concurrently treated with a stable dose of a second generation antipsychotic.

DETAILED DESCRIPTION:
The primary features of schizophrenia are characterized by positive (irrational thoughts and/or behavior) and negative symptoms. Negative symptoms are the gross absence of normal behavior and emotions, and usually include a general lack of engagement, social withdrawal, and loss of goal-directed behavior.

Negative symptoms may strongly affect daytime activities and quality of life. The effects of currently available antipsychotics on negative symptoms are not satisfactory and leave much room for improvement. MK-8435 (Org 25935) is an investigational drug that may help to correct the above characteristics of schizophrenia by facilitating the messenger function of an amino acid in the brain, called glutamate. Preliminary data suggest that lowered glutamate levels in schizophrenia are associated with a failure to activate relevant areas in the forebrain and with prominent negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Is diagnosed with non-first episode schizophrenia meeting Diagnostic and Statistical Manual (Version IV) criteria
* Is receiving stable treatment with one of the following SGA: aripiprazole, olanzapine, quetiapine, risperidone, or ziprasidone
* Is in the non-acute phase of illness and clinically stable for 3 months prior to study start as demonstrated by: treatment with current SGA or at least 12 weeks prior to study start; no increase in the level of psychiatric care due to worsening symptoms for at least 12 weeks prior to study start; and no dose change of SGA or change in medication to treat the symptoms of schizophrenia for 4 weeks prior to study start
* Has a score ≥4 on 3 or more of the following Positive and Negative Symptoms Scale (PANSS) negative subscale items at study start: blunted affect, emotional withdrawal, poor rapport, passive social withdrawal, lack of spontaneity, motor retardation, and active social avoidance
* Has an overall PANSS negative subscale score > 20

Exclusion Criteria:

* Has an overall PANSS positive subscale score ≥20
* Has a score ≥5 on 2 or more of the following PANSS positive subscale items at study start: delusions, hallucinatory behavior, excitement, grandiosity, or suspiciousness/persecution
* Has a score ≥9 on the modified InterSePT Scale for Suicidal Thinking
* Has a score ≥9 on the Calgary Depression Scale for Schizophrenia
* Has a score ≥3 on the clinical global impression of Parkinsonism of the abbreviated Extrapyramidal Symptom Rating Scale
* Has untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, cardiovascular, hematological, immunological or cerebrovascular disease, malignancy, or other chronic and/or degenerative process
* Has a history of seizure disorder beyond childhood or is taking any anticonvulsants to prevent seizures
* Has a diagnosis of mental retardation or organic brain syndrome
* Has a clinically relevant visual disturbance, such as cataract, color blindness, macular degeneration, glaucoma, or retinal disease
* Has a concurrent diagnosis of substance dependence other than nicotine or caffeine dependence in the past 6 months prior to study start
* Has a positive result on the urine alcohol/drug screen for alcohol or illicit drugs
* Is pregnant or breastfeeding
* Is being treated with high doses of benzodiazepines (>4 mg per day lorazepam or equivalent)
* Has an imminent risk of self-harm or harm to others
* Has been treated with clozapine in the past 6 months prior to study start
* Has been treated with lithium, valproate, lamotrigine, pregabalin, gabapentin, or carbamazepine in the past 12 weeks prior to study start
* Has started treatment or has had a dose change of an (additional) antipsychotic, antidepressant,hypnotic or anxiolytic in the past 4 weeks prior to study start
* Has had no demonstrated benefit of antipsychotic treatment within the previous five years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2007-04-10 (Actual); Primary Completion 2008-10-24 (Actual); Study Completion 2008-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Schoemaker JH, Jansen WT, Schipper J, Szegedi A. The selective glycine uptake inhibitor org 25935 as an adjunctive treatment to atypical antipsychotics in predominant persistent negative symptoms of schizophrenia: results from the GIANT trial. J Clin Psychopharmacol. 2014 Apr;34(2):190-8. doi: 10.1097/JCP.0000000000000073. PMID 24525661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were maintained on a stable dose of Second Generation Antipsychotic (SGA) and received add-on therapy with MK-8435 (Org 25935). 215 participants were randomized and 214 participants were treated. There was no stratification for SGA treatment.
Groups:
- MK-8435 (Org 25935) 8-16 mg Per Day: Participants were maintained on a stable dose of Second Generation Antipsychotic (SGA) and received 4-8 mg MK-8435 (Org 25935) twice a day (BID), in the morning and the evening, as add-on treatment for up to 87 days. The dose of MK-8435 (Org 25935) was titrated upward or downward within the specified dose range, as needed, up to Day 42 of the study. The dose remained stable after Day 42 for the remainder of the study.
- MK-8435 (Org 25935) 24-32 mg Per Day: Participants were maintained on a stable dose of SGA and received 12-16 mg MK-8435 (Org 25935) BID, in the morning and the evening, as add-on treatment for up to 87 days. The dose of MK-8435 (Org 25935) was titrated upward or downward within the specified dose range, as needed, up to Day 42 of the study. The dose remained stable after Day 42 for the remainder of the study.
- Placebo: Participants were maintained on a stable dose of SGA and received matching placebo for MK-8435 (Org 25935) BID, in the morning and the evening, as add-on treatment for up to 87 days.
Period: Overall Study
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Started | 72 | 73 | 70
Treated | 71 | 73 | 70
Completed | 61 | 65 | 61
Not Completed | 11 | 8 | 9
Not completed — Use of Excluded Medication | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 4
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Worsening of Disease | 2 | 1 | 2
Not completed — Inclusion/Exclusion Criteria | 1 | 0 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo | Total
Number analyzed (Participants) | 72 | 73 | 70 | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (10.1) | 38.8 (11.0) | 38.1 (10.5) | 38.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 24 | 82
  Male | 41 | 46 | 46 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Scale for the Assessment of Negative Symptoms (SANS 1-22 Composite Score) at Week 12
Description: SANS was a 25-item clinician-rated instrument for assessing the negative symptoms of schizophrenia. SANS 1-22 Composite Score consisted of the SANS 25 scale minus the last 3 questions (attention items). The remaining non-attention items (affective flattening, alogia, avolition-apathy, and anhedonia-asociality) comprised the SANS 1-22 Composite Score. For each item, symptom severity was rated on a 6-point scale, from 0=absent to 5=severe. The SANS 1-22 Composite Score had a total scoring range of 0 to 110. Higher scores indicated more impairment. The SANS 1-22 Composite Score was reported using data from the adjusted site rater. A negative change from baseline indicated an improvement in symptoms.
Time Frame: Baseline and Week 12
Population: All randomized participants who received either MK-8435 (Org 25935) or placebo and who completed at least 8 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | -13.50 (12.58) | -10.91 (11.85) | -11.21 (11.28)
Statistical Analysis 1: Comparison: MK-8435 (Org 25935) 8-16 mg Per Day vs Placebo; Comparison of Mean Change in Baseline: Least Squared Estimates with Statistical Inference; Test type: Superiority or Other; p = 0.267, ANCOVA; ANCOVA model with the baseline value as covariate and with treatment group and center as fixed factors; Mean Change From Baseline = -2.26, 95% CI 2-sided [-6.25 to 1.74]
Statistical Analysis 2: Comparison: MK-8435 (Org 25935) 24-32 mg Per Day vs Placebo; Comparison of Mean Change in Baseline: Least Squared Estimates with Statistical Inference; Test type: Superiority or Other; p = 0.966, ANCOVA; ANCOVA model with the baseline value as covariate and with treatment group and center as fixed factors; Mean Change From Baseline = -0.08, 95% CI 2-sided [-3.91 to 3.74]

2. Secondary Outcome: Change From Baseline in Total Score of Positive and Negative Syndrome Scale (PANSS) for Schizophrenia at Week 12
Description: PANSS was a 30-item clinician-rated instrument used for assessing the positive, negative, and general psychopathology symptoms of schizophrenia. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme, with a total scoring range of 30 to 210. Higher scores indicated more impairment. A negative change from baseline indicated an improvement in symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | -11.84 (10.34) | -10.69 (10.40) | -9.73 (11.23)

3. Secondary Outcome: Change From Baseline in the Calgary Depression Scale for Schizophrenia (CDSS) at Week 12
Description: CDSS was a 9-item clinician-rated instrument used to evaluate depression in participants who have schizophrenia. For each item, symptom severity was rated on a 4-point scale, from 0=absent to 3=severe, with a total scoring range of 0 to 27. Higher scores indicated more impairment. A negative change from baseline indicated an improvement in symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | -0.95 (1.88) | -0.76 (1.88) | -0.56 (2.67)

4. Secondary Outcome: Change From Baseline in Perception of Emotions Score at Week 12
Description: Perception of emotion was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery. The participant identified different emotional states (happy, sad, angry, and calm [neutral]) presented in pictures of faces by choosing the appropriate word for the emotion. The raw score was the sum of correct responses minus errors. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 1.42 (4.18) | 1.55 (4.35) | -0.80 (5.91)

5. Secondary Outcome: Change From Baseline in Non-Verbal Reasoning Score at Week 12
Description: Non-verbal reasoning was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery. The participant solved 15 visual analogies composed of geometric 2x2, 3x3, or 4x4 puzzles by choosing the most appropriate geometric figure that solved the matrix. The raw score was the sum of correct responses minus errors. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 0.65 (4.30) | 0.66 (3.95) | 0.78 (4.68)

6. Secondary Outcome: Change From Baseline in Verbal Memory Score at Week 12
Description: Verbal memory was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery. The participant remembered 15 words within a field of 15 distractors immediately and after a twenty minute delay. The raw score was the sum of correct responses. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | -0.76 (7.61) | 0.41 (7.85) | -0.78 (8.60)

7. Secondary Outcome: Change From Baseline in Visual Memory Score at Week 12
Description: Visual memory was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery. The participant remembered 15 geometric figures within a field of 15 distractors immediately and after a twenty minute delay. The raw score was the sum of correct responses. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sore on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Sore on a Scale | -0.35 (4.98) | -1.73 (6.20) | -1.34 (6.59)

8. Secondary Outcome: Change From Baseline in Speed of Complex Information Processing Score at Week 12
Description: Speed of complex information processing was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery-Symbol-digit Coding Test. The participant linked numbers to digits. The test consisted of serial presentations of screens, each containing a bank of 8 symbols above and 8 empty boxes below. The participant typed the number that corresponded to the symbol highlighted. The raw score was the processing time in milliseconds. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 5.62 (8.53) | 5.73 (13.21) | 5.17 (12.94)

9. Secondary Outcome: Change From Baseline in Working Memory Score at Week 12
Description: Working memory was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery-4-Part Continuous Performance Test. The participant was presented with targets and remembered target presentation sequencing in order to respond to the directions. Only Part 4 of the 4 Part Continuous Performance Test contributed towards the working memory score. The raw score was the sum of correct responses minus errors. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 0.96 (4.62) | 0.37 (4.75) | 0.82 (6.72)

10. Secondary Outcome: Change From Baseline in Sustained Attention Score at Week 12
Description: Sustained attention was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery-4-Part Continuous Performance Test. The participant was asked to identify a target shape/color when presented with a battery of different geometric shapes/colors. Only Parts 2 to 4 of the 4 Part Continuous Performance Test contributed towards the sustained attention score. The raw score was the sum of correct responses minus errors. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 0.96 (10.76) | 3.81 (11.14) | 1.95 (15.88)

11. Secondary Outcome: Change From Baseline in Executive Functioning Score at Week 12
Description: Executive functioning was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery-Shifting Attention Test. The participant matched geometric shapes either by shape or color. The raw score was the sum of correct responses minus errors. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: All randomized participants who received ≥1 dose of study therapy and completed at least 8 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | 10.16 (19.55) | 9.33 (20.09) | 12.57 (23.26)

12. Secondary Outcome: Change From Baseline in Composite Memory Score at Week 12
Description: Composite memory was a composite of verbal memory and visual memory and was measured by computer using the CNS-Vital Signs Neurocognitive Test Battery. The raw score was the sum of correct responses. The standard scores were normalized from raw scores and presented an age-matched score relative to a normative comparison database. Higher scores were better.
Time Frame: Baseline and Week 12
Population: All randomized participants who received ≥1 dose of study therapy and completed at least 8 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 62 | 67 | 62
Score on a Scale | -1.26 (10.64) | -1.32 (11.61) | -2.12 (12.35)

13. Secondary Outcome: Change From Baseline in Extrapyramidal Symptoms Rating Scale Score at Week 12
Description: The abbreviated Extrapyramidal Symptoms Rating Scale (ESRS-A) was a sum of the severity rating of a 24-item instrument assessing four types of movement disorders: parkinsonism, dystonia, dyskinesia, and akathisia. Each item was rated on a 7-point scale, from 0=absent to 6=severe. Higher scores indicated more impairment. A negative change from baseline indicated an improvement.
Time Frame: Baseline and Week 12
Population: All randomized participants who received ≥1 dose of study therapy.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Number analyzed (Participants) | 71 | 73 | 70
Score on a Scale | -0.8 (2.2) | -0.3 (1.2) | -1.0 (3.4)

ADVERSE EVENTS:
Time Frame: From treatment Day1 through follow-up (up to 120 days)
Description: AEs were reported for all randomized participants who received ≥1 dose of study therapy for both the treatment and follow-up periods.
Arm/Group | MK-8435 (Org 25935) 8-16 mg Per Day | MK-8435 (Org 25935) 24-32 mg Per Day | Placebo
Serious Adverse Events (participants affected / at risk) | 2/71 | 2/73 | 1/70
Other Adverse Events (participants affected / at risk) | 15/71 | 26/73 | 17/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8435 (Org 25935) 8-16 mg Per Day (N=71) | MK-8435 (Org 25935) 24-32 mg Per Day (N=73) | Placebo (N=70)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8435 (Org 25935) 8-16 mg Per Day (N=71) | MK-8435 (Org 25935) 24-32 mg Per Day (N=73) | Placebo (N=70)
Tachycardia (Cardiac disorders) | 2 (2) | 4 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 7 (10) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (6) | 7 (7)
Somnolence (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (7) | 5 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the sponsor at least six weeks ahead of estimated publication or presentation, for written consent. The sponsor shall have the right to make its consent of information conditional upon proper representation of the interpretation of both the sponsor and the investigator(s) in the discussion of the data in such communications.